CLINICAL TRIAL: NCT03433716
Title: Ultrasound-guided Percutaneous Neuromodulation in Patients With Lateral Epicondylalgia: a Pilot Randomized Clinical Trial
Brief Title: Neuromodulation in Lateral Elbow Pain
Acronym: PNM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blanca de la Cruz Torres (Other)
Responsible Party: Sponsor-Investigator, Blanca de la Cruz Torres, PT, PhD, University of Seville
Organization: University of Seville (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PNM
Record Dates: First submitted 2018-02-01; First posted 2018-02-15 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Lateral Epicondylitis
Keywords: Percutaneous Neuromodulation, radial nerve, pain
MeSH Terms: conditions — Tennis Elbow; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNM group (Experimental): Subjects were treated for 3 weeks, once a week. Specifically, this consisted in the application of a square wave biphasic electrical current, with 10Hz frequency, a 250µs pulse width, and the maximal tolerable intensity to cause an exacerbated muscle contraction for a total of 1.5 mins, according to the protocol by Valera and Minaya. The subjects were seated while their arms were supported by an arm rest, forearms pronated and elbows moderately flexed. The radial nerve was located at 4cm proximal to the tip of the lateral epicondyle of humerus using an ultrasound machine (cross-section), subsequently, an acupuncture needle (0.30mm x 30mm) was inserted in a short axis approach, perpendicular to the surface of the skin, until the perineurium of the radial nerve (in close proximity).
  Interventions: Other: Ultrasound-guided Percutaneous Neuromodulation
- Control group (No Intervention): the subects of the control group received no any treatment

INTERVENTIONS:
Other: Ultrasound-guided Percutaneous Neuromodulation — It's a new intervention of sport physiotherapy. It´s an invasive technique. It is necessary an ultrasound
  Arms: PNM group

SUMMARY:
Lateral epicondylitis (LE), also known as tennis elbow, refers to a painful condition at or around the lateral epicondyle of the humerus and common extensor tendon (CET) that is aggravated by dorsiflexion and/or supination of the wrist against resistance. Lateral epicondylitis is one of the most common injuries of the elbow, affecting 1-3% of the population.

Therefore, determining an effective intervention that helps manage the condition and lessens the financial burden is important. Passive physical modalities, including electrotherapy and orthotic devices, are common treatments for the management of elbow pain. Passive physical modalities are physical treatments involving a device that does not require active participation by the patient. In a systematic review, 2017, Dion et al examined the effectiveness of passive physical modalities for the treatment of soft tissue injuries of the elbow, but little evidence exists to support or refute their use.

Clinically, an invasive technique has appeared, known as Ultrasound-guided Percutaneous Neuromodulation (PNM). This minimally invasive intervention consists in the applicacion of a percutaneous electrical stimulation (PES) through an acupuncture needle-like electrode that is placed in close proximity to the nerve or motor point of the muscle with ultrasound guidance. At the clinical level, the PES is always used with the therapeutic aim of relieving chronic pain and neuropathic pain. Similarly, in sports, PES is used with the aim of improving muscular activity. Therefore, according to the characteristics and the therapeutic benefits of this technique, further research is needed to discover multiple clinical indications.

The aim of this pilot study was to examine the effects of a percutaneous neuromodulation intervention in patients with unilateral refractory lateral epicondylitis. Findings from this study may provide further evidence for the relevance of neural tissues in determining the elbow pain and may indicate effects of US-guided NMP technique on the rehabilitation and/or prevention of in patients with unilateral refractory LE.

ELIGIBILITY:
Inclusion Criteria:

* Presence of pain in the elbow region at least for three months
* Flares with activity
* Tenderness at or within 2cm of the lateral humeral epicondyle on resisted extension of the wrist and/or the third finger.

Exclusion Criteria:

* Participants who had constant or radicular pain
* Any previous surgery or acute trauma in the upper extremity.
* Elbow deformity
* Bilateral symptoms
* Clinical or electrophysiological findings referable to peripheral nerve (ulnar and median) disease and

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-06 (Actual); Primary Completion 2018-05-06 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
average pain at palpation | Baseline and up to 1 month
  Numerical rating scale (NRS) (0, points; 10, maximum points).

SECONDARY OUTCOMES:
Patient-Rated Tennis Elbow Evaluation (PRTEE) | Baseline and up to 1 month
  Pain and functional ability
radial nerve cross-sectional area (CSA) | Baseline and up to 1 month
  Cross-sectional area was measure at 4cm proximal to the tip of the lateral epicondyle of humerus
Strengt-Duration (SD) curves | Baseline and up to 1 month
  chronaxie and accommodation index

CONTACTS AND LOCATIONS:
Overall Officials: BLANCA DE LA CRUZ, DR, Principal Investigator — University of Seville
Locations (1):
- Blanca de La Cruz Torres, Seville, Spain

IPD SHARING:
Plan to Share IPD: Undecided